CLINICAL TRIAL: NCT07152639
Title: Phase III Clinical Trial to Evaluate the Efficacy and Safety of Recombinant Mycobacterium Tuberculosis Fusion Protein (EEC) for the Diagnosis of Mycobacterium Tuberculosis Infection in People Aged 3 Years and Above
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of EEC for the Diagnosis of Mycobacterium Tuberculosis Infection in People Aged 3 Years and Above
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chengdu CoenBiotech Co., Ltd (Industry)
Collaborators: Beijing Chest Hospital, Capital Medical University (Other); Wuhan Pulmonary Hospital (Other); Changsha Central Hospital (Other); The First Affiliated Hospital of Xinxiang Medical College (Other); LiuZhou People's Hospital (Other); Wuhan Central Hospital (Other); Yichang Central People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: KN-EEC-III
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Community-dwelling population aged 3 - 64 years old (Experimental): 415 Community-dwelling population subjects's left and right arms were randomly assigned to receive a single intradermal injection of 0.1 ml of the test drug (EEC 5 μg /ml ) and the control drug (EC); all subjects were intradermally injected into the middle and lower 1/3 of the volar side of the forearm using the Mantoux method. injection. The time between skin tests on the left and right arms must be at least 30 minutes (skin test on the left arm first, then on the right arm). The follow-up visit observation point is based on the completion time of the second dose of injection.
  Interventions: Biological: 5μg/ml EEC; Biological: 5 unit（U） EC; Diagnostic Test: IGRA
- Community-dwelling population aged above 18 years old (Experimental): 334 Community-dwelling population subjects's left and right arms were randomly assigned to receive a single intradermal injection of 0.1 ml of the test drug (EEC 5 μg /ml ) and the control drug (TB-PPD); all subjects were intradermally injected into the middle and lower 1/3 of the volar side of the forearm using the Mantoux method. injection. The time between skin tests on the left and right arms must be at least 30 minutes (skin test on the left arm first, then on the right arm). The follow-up visit observation point is based on the completion time of the second dose of injection.
  Interventions: Biological: 5μg/ml EEC; Biological: 5 IU TB-PPD; Diagnostic Test: IGRA
- BCG vaccination subjects in triple-negative population (Experimental): Cohort 2 is a healthy group of participants (i.e., triple-negative people) whose test results (including EEC and TB-PPD) and IGRA are negative in both arms after the first skin test. 80 triple-negative people are planned to be included.
  If they meet the eligibility criteria for BCG vaccination, they will be vaccinated with BCG within 3 weeks after the first skin test, and the second skin test will be conducted again 12 weeks after vaccination.
  During the second skin test, participants will be randomly injected with a single intradermal injection of 0.1 ml of the test drugs EEC and TB-PPD in each arm.
  Interventions: Biological: 5μg/ml EEC; Biological: 5 IU TB-PPD; Diagnostic Test: IGRA
- TB subjects in 3-64 years old (Experimental): 300 TB subjects's left and right arms were randomly assigned to receive a single intradermal injection of 0.1 ml of the test drug (EEC 5 μg /ml ) and the control drug (EC); all subjects were intradermally injected into the middle and lower 1/3 of the volar side of the forearm using the Mantoux method. injection. The time between skin tests on the left and right arms must be at least 30 minutes (skin test on the left arm first, then on the right arm). The follow-up visit observation point is based on the completion time of the second dose of injection.
  Interventions: Biological: 5μg/ml EEC; Biological: 5 unit（U） EC; Diagnostic Test: IGRA
- TB subjects above 65 years old (Experimental): 235 TB subjects's left and right arms were randomly assigned to receive a single intradermal injection of 0.1 ml of the test drug (EEC 5 μg /ml ) and the control drug (TB-PPD); all subjects were intradermally injected into the middle and lower 1/3 of the volar side of the forearm using the Mantoux method. injection. The time between skin tests on the left and right arms must be at least 30 minutes (skin test on the left arm first, then on the right arm). The follow-up visit observation point is based on the completion time of the second dose of injection.
  Interventions: Biological: 5μg/ml EEC; Biological: 5 IU TB-PPD; Diagnostic Test: IGRA
- non-TB subjects with lung disease in 18-65 years old (Experimental): 300 non-TB subjects with lung disease left and right arms were randomly assigned to receive a single intradermal injection of 0.1 ml of the test drug (EEC 5 μg /ml ) and the control drug (EEC); all subjects were intradermally injected into the middle and lower 1/3 of the volar side of the forearm using the Mantoux method. injection. The time between skin tests on the left and right arms must be at least 30 minutes (skin test on the left arm first, then on the right arm). The follow-up visit observation point is based on the completion time of the second dose of injection.
  Interventions: Biological: 5μg/ml EEC; Biological: 5 unit（U） EC; Diagnostic Test: IGRA
- non-TB subjects with lung disease above 65 years old (Experimental): 200 non-TB subjects with lung disease left and right arms were randomly assigned to receive a single intradermal injection of 0.1 ml of the test drug (EEC 5 μg /ml ) and the control drug (TB-PPD); all subjects were intradermally injected into the middle and lower 1/3 of the volar side of the forearm using the Mantoux method. injection. The time between skin tests on the left and right arms must be at least 30 minutes (skin test on the left arm first, then on the right arm). The follow-up visit observation point is based on the completion time of the second dose of injection.
  Interventions: Biological: 5μg/ml EEC; Biological: 5 IU TB-PPD; Diagnostic Test: IGRA

INTERVENTIONS:
Biological: 5μg/ml EEC — 0.1ml, one time, containing high dose 5μg/ml of active ingredients
Biological: 5 unit（U） EC — 0.1 ml , one time, containing 5U of active ingredients
  Arms: Community-dwelling population aged 3 - 64 years old; TB subjects in 3-64 years old; non-TB subjects with lung disease in 18-65 years old
Biological: 5 IU TB-PPD — 0.1 ml , one time, containing 5IU of active ingredients
  Arms: BCG vaccination subjects in triple-negative population; Community-dwelling population aged above 18 years old; TB subjects above 65 years old; non-TB subjects with lung disease above 65 years old
Diagnostic Test: IGRA — 96-well/plate x 2 plates; 100 tubes/box x 1 box

SUMMARY:
This study is a randomized, blinded, active-controlled clinical trial to evaluate the effectiveness and safety of EEC in the diagnosis of Mycobacterium tuberculosis infection in people aged 3 years and above.

Methods: In study 1, the marketed recombinant Mycobacterium tuberculosis fusion protein (EC) was used as a control drug in people aged 3 to 64 years. The sensitivity of EEC in participants with tuberculosis and the specificity in healthy participants and patients with non-tuberculous lung diseases were evaluated compared with recombinant Mycobacterium tuberculosis fusion protein (EC). The clinical positivity criteria of EEC were verified, and the consistency of the two detection methods, as well as the safety of EEC, were evaluated.

Study 2: Triple-negative people aged 18 and above (negative in EEC, TB-PPD, and IGRA tests) were screened out from the community population and vaccinated with BCG. EEC and TB-PPD double-arm skin tests were performed 12 weeks after vaccination to evaluate whether there was a significant difference in the negative rate of EEC compared with TB-PPD after BCG vaccination in the triple-negative population.

Study 3: A multicenter, positive-controlled, non-inferiority trial design was used for people aged 65 years and above, and the research hypothesis was independently tested to verify the non-inferiority of the sensitivity of this product in tuberculosis patients in this age group compared with IGRA and TB-PPD, as well as the consistency of the diagnostic results of IGRA with non-tuberculous lung diseases and the general community population. At the same time, attention was paid to and analysis of the specificity and safety of EEC in people aged 65 years and above.

DETAILED DESCRIPTION:
This study is a randomized, blinded, active-controlled clinical trial to evaluate the effectiveness and safety of EEC in the diagnosis of Mycobacterium tuberculosis infection in people aged 3 years and above.

Study 1: The marketed recombinant tuberculosis fusion protein (EC) was used as a control drug in the population aged 3-64 years: This clinical trial adopted a multicenter, randomized, positive-controlled, blinded, homologous double-arm, non-inferiority trial design in the population aged 3-64 years, aiming to evaluate the sensitivity of EEC compared with recombinant tuberculosis fusion protein (EC) in participants with tuberculosis, the specificity in healthy participants and patients with non-tuberculous lung diseases, verify the clinical positive judgment criteria of EEC, and evaluate the consistency of the two detection methods of EEC and EC and the safety of EEC.

Study 2: The marketed tuberculin purified protein derivative (TB-PPD) was used as a control drug in the triple-negative population aged 18 years and above:

The triple-negative population (EEC, TB-PPD, and IGRA tests were all negative) was screened out from the community population and vaccinated with BCG. After 12 weeks of vaccination, EEC and TB-PPD were tested in the same arm to evaluate the significant difference in the negative rate of EEC compared with TB-PPD in the triple-negative population after BCG vaccination.

Study 3: TB-PPD and in vitro diagnostic reagent IGRA were used as controls for people aged 65 and above:

For people aged 65 and above, a multicenter, positive control, non-inferiority trial design was used to conduct a separate study hypothesis to verify the non-inferiority of the sensitivity of this product in tuberculosis patients in this age group compared with IGRA and TB-PPD, as well as the consistency of the diagnostic results of non-tuberculous lung diseases and the general community population with IGRA. At the same time, the specificity and safety of EEC in people aged over 65 were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* For the general community population

  1. Age 3 years and above at the time of enrollment, regardless of gender;
  2. The individual and/or guardian agree to participate in this trial and sign the informed consent form;
  3. The individual and/or guardian can comply with the requirements of the clinical trial protocol to participate/accompany the participants to participate in follow-up;
  4. No history of tuberculosis (including intrapulmonary and extrapulmonary tuberculosis) after medical history inquiry;
  5. No clinical symptoms of tuberculosis poisoning. Tuberculosis poisoning symptoms refer to obvious systemic symptoms such as fatigue, low fever in the afternoon, loss of appetite, night sweats, etc. in addition to local symptoms such as cough, chest pain, and chest tightness. Women may have endocrine system disorders, such as irregular menstruation, amenorrhea, etc.;
  6. Inclusion criteria for triple-negative population: People with negative results of the first skin test on both arms and IGRA test results (i.e., negative results of EEC, TB-PPD, and IGRA tests).
* For Patients with tuberculosis (including pulmonary tuberculosis)

  1. Age 3 years and above at the time of enrollment, regardless of gender;
  2. Participants aged ≥18 years were diagnosed with tuberculosis/pulmonary tuberculosis according to the diagnostic standard "Standard Tuberculosis Classification of the Health Industry of the People's Republic of China WS196-2017" issued by the health and health authorities of the State Council (recognizing the diagnosis made by comprehensive clinical analysis); participants aged 3-17 years were diagnosed with tuberculosis according to the "Expert Consensus on Diagnosis of Childhood Pulmonary Tuberculosis (2022 Edition)" formulated by the Children's Tuberculosis Professional Committee of the Tuberculosis Branch of the Chinese Medical Association. Including pulmonary tuberculosis and extrapulmonary tuberculosis, of which pulmonary tuberculosis includes bacteria-negative/bacteria-positive pulmonary tuberculosis and primary/relapsed pulmonary tuberculosis; patients with both pulmonary tuberculosis and extrapulmonary tuberculosis can be included and classified as pulmonary tuberculosis;
  3. The individual and/or guardian agree to participate in this trial and sign the informed consent form;
  4. The individual and/or guardian can comply with the requirements of the clinical trial protocol to participate in follow-up.

For Patients with non-tuberculous lung disease

1. Patients with a clear clinical diagnosis of non-tuberculous lung disease, and clinical physicians can exclude pulmonary tuberculosis and extrapulmonary tuberculosis based on the patient's clinical manifestations, imaging and laboratory tests, including pneumonia, lung cancer, bronchitis, bronchiectasis, non-tuberculous mycobacterial disease, chronic obstructive pulmonary disease, etc.;
2. Aged 3 years and above at the time of enrollment, regardless of gender;
3. The individual and/or guardian agree to participate in this trial and sign the informed consent form;
4. The individual or guardian can comply with the requirements of the clinical trial protocol to participate in follow-up.

Exclusion Criteria:

- For the general community population

1. Those with known or suspected (or high-risk) severe immune diseases, immune function damage or abnormalities (Except for human immunodeficiency virus [HIV] infection/HIV infection), including:Those who received immunosuppressants (including chemotherapy) (using medium/high doses of glucocorticoids (≥20mg/d or ≥0.5mg/kg/d prednisone or equivalent other hormones), and the medication time was >14 days) or immunopotentiators within 3 days before the skin test or during the trial, and those who were evaluated by the researchers to affect the efficacy of the participants; Note: For glucocorticoid drugs: topical inhalation, nasal spray, local injection, application and other external use, as well as long-term physiological replacement therapy for systemic medication such as oral, intramuscular injection, intravenous injection or intravenous drip, there are no restrictions, such as prednisone or other equivalent doses of other drugs with a dose of <20mg/d (>5 years old) or <0.5mg/kg/d (≤5 years old), and the medication time is ≤14 days.
2. Patients with convulsions, epilepsy, history of mental illness and/or family history of mental illness (immediate relatives);
3. Patients with allergic constitution, such as those with a history of allergy to two or more drugs or foods, or those known to be allergic to the components of this drug;
4. Patients with acute infectious diseases (such as measles, whooping cough, influenza, etc.), acute conjunctivitis, acute otitis media, and extensive skin diseases;
5. Patients with acute febrile diseases; or those who have used antipyretic, analgesic and antiallergic drugs within 3 days before the skin test and who have been assessed by the researchers to be likely to affect the study evaluation;
6. Patients with severe skin infections (such as pyoderma, severe eczema, etc.);
7. Those who have used other clinical trial drugs within 3 months before the skin test (except placebo, in vitro diagnostic reagents or non-contact human devices);
8. Those who have received inactivated vaccines within 7 days before the skin test, or attenuated live vaccines within 28 days;
9. Women who are breastfeeding or pregnant, or women of childbearing age who have a positive pregnancy test before enrollment. 10) Those with a history of drug abuse;

11) Those who the researcher believes have poor compliance, past history, physical examination results that may affect the trial evaluation (such as tattoos, etc.); 12) Exclusion criteria for triple-negative population: Those with contraindications to BCG vaccination, including: ① Those with immunodeficiency or damage (such as AIDS patients); ② Those currently using immunosuppressive drugs or radiotherapy; ③ Those who are allergic to BCG; ④ Those with fever and acute infectious diseases, including active tuberculosis patients; ⑤ Severe chronic diseases (such as heart, brain, vascular diseases, chronic kidney disease).

For Patients with tuberculosis and non-tuberculous lung disease

1. Those with known or suspected (or high-risk) severe immune diseases, immune function damage or abnormalities (Except for human immunodeficiency virus [HIV] infection/HIV infection), including: Those who are receiving immunosuppressants (including chemotherapy) (using medium/high doses of glucocorticoids (≥20mg/d or ≥0.5mg/kg/d), medication time>14 days) or immunoenhancers within 3 days before the skin test or during the trial, and those who are assessed by the researchers to affect the efficacy of the participants; Note: For glucocorticoid drugs: topical inhalation, nasal spray, local injection, application and other external use, as well as long-term physiological replacement therapy for systemic medication such as oral, intramuscular injection, intravenous injection or intravenous drip, there are no restrictions, such as prednisone or other equivalent doses of other drugs at a dose of <20mg/d (>5 years old) or <0.5mg/kg/d (≤5 years old), medication time ≤14 days.
2. Patients with convulsions, epilepsy, history of mental illness and/or family history of mental illness (immediate relatives);
3. Patients with allergic constitution, such as those with a history of allergy to two or more drugs or foods, or those known to be allergic to the components of this drug;
4. Patients with acute infectious diseases (such as measles, whooping cough, influenza, etc.), acute conjunctivitis, acute otitis media, and extensive skin diseases;
5. Patients with severe skin infections (such as pyoderma, severe eczema, etc.);
6. Patients who have used other clinical trial drugs within 3 months before the skin test (except placebo, in vitro diagnostic reagents or non-human contact devices);
7. Patients who have received inactivated vaccines within 7 days before the skin test, or attenuated live vaccines within 28 days;
8. Women who are breastfeeding or pregnant, or women of childbearing age who have a positive pregnancy test before enrollment.
9. Patients with a history of drug abuse;
10. Any situation that the researcher believes has poor compliance, past history, and physical examination results may affect the trial evaluation (such as tattoos, etc.).

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1784 (Estimated)
Dates: Start 2025-08-09 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity (true positive rate) of EEC and EC detection methods in tuberculosis patients aged 3 to 64 years | 7 days after injection
  Sensitivity (also known as the true positive rate which is defined as the percentage of actual disease that is correctly judged to be diseased according to the diagnostic criteria of the test) of EEC and EC detection methods in tuberculosis patients aged 3 to 64 years
Specificity (true negative rate) of EEC and EC detection methods in patients with non-tuberculous lung diseases aged 3 to 64 years | 7 days after injection
  Specificity (also known as true negative rate which is defined as the percentage of actual disease-free patients correctly judged to be disease-free according to the diagnostic criteria of the test) of EEC and EC detection methods in patients with non-tuberculous lung diseases aged 3 to 64 years
Specificity (true negative rate) of EEC and EC for the diagnosis of Mycobacterium tuberculosis infection in healthy participants aged 3-64 years . | 7 days after injection
  Specificity (true negative rate) of EEC and EC for the diagnosis of Mycobacterium tuberculosis infection in healthy participants aged 3-64 years (with no abnormal imaging, negative IGRA test results, and no symptoms/signs of tuberculosis)
Negative rate of EEC test drug and TB-PPD control drug in BCG-vaccinated population in triple-negative population | 7 days after second injection
  Negative rate of EEC test drug and TB-PPD control drug in BCG-vaccinated population in triple-negative population（including healthy subjects with negative EEC, TB-PPD and IGRA）.
Sensitivity (true positive rate) of EEC test drug versus control IGRA and TB-PPD for assisting clinical diagnosis of tuberculosis in people aged 65 years and older with tuberculosis | 7 days after injection
  Sensitivity (also known as the true positive rate which is defined as the percentage of actual disease that is correctly judged to be diseased according to the diagnostic criteria of the test) of EEC test drug versus control IGRA and TB-PPD for assisting clinical diagnosis of tuberculosis in people aged 65 years and older with tuberculosis
To evaluate the consistency (accordance rate) of the diagnostic results of EEC and IGRA in non-tuberculous lung diseases in the general community population aged 65 years and above | 7 days after injection
  The consistency rate of EC, EEC and IGRA detection reagents which is defined as the pairwise KAPPA values of the three detection methods in different dose groups among healthy people and patients with non-tuberculosis pulmonary disease( the Kappa values of the three detection methods in different dose groups were calculated respectively ).

SECONDARY OUTCOMES:
Verify the ROC curve and area under the curve (AUC) of EEC, and verify the optimal diagnostic threshold, time range, and specific reaction type (redness or induration) of the test drug | 7 days after injection
To evaluate the consistency of skin test results (positive detection rate and negative detection rate) between EEC and EC in the general community population, TB patients and patients with non-tuberculous lung diseases | 7 days after injection
Evaluate the positive rate of skin test results of EEC and TB-PPD in the general community population | 7 days after injection
The incidence of adverse events (AEs) and serious adverse events (SAEs) in EEC during the trial | 7 days after injection
  Safety endpoint including: incidence of adverse events at injection and non-injection sites within 7 days after skin test; abnormal incidence of laboratory indicators (blood routine, blood biochemistry,) at 7 days after skin test; abnormal incidence of vital signs within 7 days after skin test; incidence of serious adverse events after skin test during the study period.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Beijing Chest Hospital, Beijing, Beijing Municipality
  - Changsha Center Hospital, Hunan, Changsha
  - LiuZhou People's Hospital, Liuchow, Guangxi
  - The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan
  - Wuhan Pulmonary Hospital, Wuhan, Hubei
  - Wuhan Central Hospital, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Public health clinical center of chengdu, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided